CLINICAL TRIAL: NCT02425566
Title: Role of Sympathetic Activity and Splanchnic Capacitance in Hypertension
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 141218
Record Dates: First submitted 2015-04-10; First posted 2015-04-24 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: autonomic nervous system; hypertension; ganglionic blocker; trimethaphan; splanchnic circulation; capacitance
MeSH Terms: conditions — Hypertension | interventions — Trimethaphan; trimethaphan camsylate; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Study day with trimethaphan (Experimental): After baseline measurements, autonomic blockade will be induced by continuous intravenous infusion of trimethaphan starting at 0.5-1.0 mg/min and increasing by 1.0 mg/min every 2 to 6 minutes up to an infusion rate of 5 mg/min.
  Interventions: Drug: Trimethaphan
- Radionuclide Study day with nitroglycerin (Experimental): Sublingual nitroglycerin (0.3-0.6 mg) will be given after baseline measurements. Outcome measurements will be repeated within 10 min after the nitroglycerin has dissolved
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Trimethaphan — Trimethaphan is a Nn-nicotinic receptor antagonist that blocks sympathetic and parasympathetic transmission at the level of the autonomic ganglia. It will be administered as an acute intravenous infusion with doses ranging from 0.5 to 5.0 mg/min.
  Other Names: Trimethaphan Camsylate
  Arms: Study day with trimethaphan
Drug: Nitroglycerin — Sublingual nitroglycerin (0.3-0.6 mg) will be given after baseline measurements.
  Other Names: Nitroglycerin sublingual, nitrostat
  Arms: Radionuclide Study day with nitroglycerin

SUMMARY:
The purpose of this study is to better understand the role of the abdominal veins (splanchnic capacitance) and the sympathetic nervous system in human hypertension. The investigators will test the hypothesis that constriction of abdominal veins due to sympathetic activation contributes to human hypertension. Splanchnic capacitance will be assessed in normotensive and hypertensive subjects at baseline and during acute blockade of the autonomic nervous system.

DETAILED DESCRIPTION:
The splanchnic circulation contains a highly compliant venous bed which normally stores ~25% of the blood volume, and receives up to 25% of the resting cardiac output. It is highly innervated by the sympathetic nervous system, and this neural regulation results in large volume shifts that modulate blood pressure (BP). The splanchnic circulation may play a role in hypertension as suggested by studies showing that surgical splanchnic denervation effectively lowered BP in hypertensive subjects without affecting renal function. Recently, studies in animal models have shown that splanchnic sympathetic activation, particularly to capacitance vessels, was critical to the development of hypertension. The clinical translation of these findings to human hypertension has lagged behind because of limitations in previously available experimental approaches. The investigators propose to use splanchnic radionuclide plethysmography and sympathetic withdrawal with the ganglionic blocker trimethaphan to overcome these limitations.

Several studies have shown that sympathetic activity contributes to hypertension. Accordingly, our previous studies showed that sympathetic withdrawal with the ganglionic blocker trimethaphan resulted in normalization of BP in hypertensive subjects. Interestingly, this was caused mainly by a fall in stroke volume, rather than a decrease in arterial vascular resistance suggesting that decreased venous return may play a major role, and that a sympathetically mediated contraction of splanchnic capacitance contributes to the maintenance of hypertension.

The investigators hypothesize that the decrease in BP induced by autonomic blockade with trimethaphan results from an increase in splanchnic capacitance leading to a reduction in venous return. To test this hypothesis, the investigators will compare the effect of sympathetic withdrawal on splanchnic capacitance between hypertensive and normotensive subjects. Splanchnic venous capacitance will be measured by radionuclide plethysmography. Abdominal blood volumes will be measured using labeled red cells with technetium-99 while applying different levels of continuous positive airway pressure.

In addition, the investigators will assess whether changes in splanchnic capacitance measured by bioimpedance are similar to those measured by radionuclide imaging. For this purpose, the investigators will compare the effects of nitroglycerin on splanchnic capacitance measured by the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Lean and obese, male and female subjects of all races between 18 and 65 years of age.
* Normotensive and hypertensive subjects will be enrolled. Hypertension will be defined as a systolic BP ≥140 mm Hg and/or a diastolic BP ≥ 90 mm Hg, taken in the seated position in at least 2 separate occasions. All subjects will be otherwise normal volunteers.
* Subjects able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Subjects with morbid obesity (BMI > 40 kg/m2).
* Subjects with any chronic disease (other than hypertension) including diabetes, cardiovascular disease, history of smoking, or if they take any medication that have known effects autonomic functions, or other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.
* Current smokers or history of heavy smoking (>2 packs/day)
* Lean normotensive subjects will be excluded if they have a strong family history of hypertension (both parents treated or diagnosed), diagnosis of sleep apnea or a high score in the Berlin questionnaire for sleep apnea, or if they are highly trained athletes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Splanchnic venous capacitance | after 10 minutes of autonomic blockade
  The primary outcome will be the splanchnic capacitance, defined as the pressure-venous curve (P-V curve), during trimethaphan infusion adjusted for its baseline values. For analysis, the Y-intercept (volume) and the slope of the P-V relationship during autonomic blockade adjusted by their corresponding baseline values will be compared between groups.

SECONDARY OUTCOMES:
Systolic Blood Pressure | after 10 minutes of autonomic blockade
  Changes from baseline in blood pressure.
Stroke volume | after 10 minutes of autonomic blockade
  Changes from baseline in stroke volume.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Autonomic Dysfunction Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okamoto LE, Dupont WD, Biaggioni I, Kronenberg MW. Effect of nitroglycerin on splanchnic and pulmonary blood volume. J Nucl Cardiol. 2022 Dec;29(6):2952-2963. doi: 10.1007/s12350-021-02811-7. Epub 2021 Nov 2. PMID 34729682